CLINICAL TRIAL: NCT06595823
Title: Betadine Versus Saline in Swapping of Subcutaneous Tissue to Prevent Surgical Site Infection After Caesarian Section
Brief Title: Betadine Versus Saline in Swapping of Subcutaneous Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asmaa Gamal Mohamed
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2022-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Povidone-Iodine10%) (Active Comparator): About 100 patients women who underwent elective caesarian section with subcutaneous tissue irrigation with Povidone iodine 10% solution.
  Interventions: Drug: Betadine
- Group B (Saline0.9%) (Active Comparator): About 100 patients women who underwent elective caesarian section with subcutaneous tissue irrigation with normal saline0.9%
  Interventions: Drug: Betadine
- Group C (the control group) (Placebo Comparator): About 100 patients women who underwent elective caesarian section without irrigation of the subcutaneous tissue with betadine or saline.
  Interventions: Drug: Betadine

INTERVENTIONS:
Drug: Betadine — To compare between Betadine (10%) and saline (0.9%) in swapping of subcutaneous tissue for prevention of surgical site infection after primary elective caesarian section.
  Other Names: Saline

SUMMARY:
Caesarean section is an increasingly common major surgical procedure performed on women. Last decade an overall increase of the global rate of caesarean section, of up to 31.2%, was reported. The risk of maternal morbidity and mortality is higher in caesarean section than in vaginal birth; postoperative infection is a common component of morbidity. With the increase in caesarean section, it is important that the risks to the mother are minimized as far as possible.

Women who give birth by caesarean section are exposed to both endogenous (internal) and exogenous (external) sources of infection during birth. Exposure to a hospital environment places these women at risk of developing hospital-acquired infections. The rate of post-caesarean infection has been estimated to be 10 times greater than that after vaginal birth.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) estimates that 27 million surgical procedures are performed in the United States each year. The CDC's National Nosocomial Infections Surveillance system reports that surgical site infections are the third most frequently reported nosocomial infection, accounting for 14% to 16% of all such infections.

Preventing infection by properly preparing the skin before incision is thus a vital part of the overall care given to women during caesarean birth. The incidence of abdominal incisional infections following caesarean section ranges from 3% to 15%.A post-caesarean surgical site infection is a bacterial infection in the surgical incision following an abdominal birth. Women who develop a post-caesarean surgical site infection typically experience a temperature of 38.0°C (100.4°F) or higher and lower abdominal pain. Abdominal incisional abscesses that develop following caesarean birth usually cause fever on about the fourth postoperative day.

In many cases, these are preceded by uterine infection, and fever persists from the first or second postoperative day. Wound redness (erythema) and drainage may also be present. Organisms causing these infections are usually the same as those isolated from amniotic fluid at caesarean birth, but hospital-acquired pathogens may also be the cause. Some women are more likely than others to develop a post-caesarean surgical site infection.Women at increased risk include those who are obese; have diabetes or an immunosuppressive disorder (HIV infection); have chorioamnionitis (infection of the amniotic fluid and fetal membrane) during labor; anemia; or are taking corticosteroids.

Proper preparation of an incision site involves removing surface dirt and oil with a soap or detergent scrub plus applying a topical antimicrobial agent that will reduce the bacterial population to a minimal level.If prophylactic antimicrobials are given, the incidence of abdominal wound infection following cesarean delivery ranges from 2 to 10 percent depending on risk factors. Numerous good quality trials have proved that a single dose of an antimicrobial agent given at the time of cesarean delivery significantly decreases infection morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Primary Elective Cs .
* Age: 20 - 35 years old,
* elective caesarean section time from skin incision to skin closure less than 60 minute,
* Body Mass Index: 20- 30 Kg/m2.

Exclusion Criteria:

* Diabetes mellitus,
* feverish patient,
* patient using steroids for chronic illness,
* prelabour rupture of membrane,
* difference in pre and postoperative hemoglobin more than 10%,
* Patients with coagulopathies,
* mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Treatment of surgical site infections | 6 weeks after cesarean section
  Assessment of Number of Participants With Treatment of surgical site infections using Povidine Iodine or by using saline and which one is effective in Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abd El Hameed Ahmed, Professor, Study Chair — Obstetrics and Gynecology Department, Faculty of medicine, Al-Azhar University, Assuit.
Locations (1):
- Al-Azhar University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No